CLINICAL TRIAL: NCT05875116
Title: Effect of Different Therapeutic Modalities With Virtual Reality or Modified Constraint-induced Movement Therapy Compared With Usual Physical and Occupational Therapy on Motor Recovery of Paretic Limbs in Patients With Cerebrovascular Event
Brief Title: Virtual Reality Versus Constraint-induced Movement on Hemiparesis in Cerebrovascular Event
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Responsible Party: Principal Investigator, María del Carmen Rojas-Sosa, Principal Investigator, Coordinación de Investigación en Salud, Mexico
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R 2016 3702 44
Record Dates: First submitted 2023-05-03; First posted 2023-05-25 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Stroke Sequelae
Keywords: Constraint-induced movement therapy; Hemiparesis; Neurorehabilitation; Satisfaction; Stroke; Virtual Reality
MeSH Terms: conditions — Paresis; Personal Satisfaction; Stroke | interventions — Occupational Therapy

STUDY DESIGN:
Intervention Model Description: Clinical Trial Randomized Single Blind
Who Masked: Outcomes Assessor
Masking Description: The evaluators were blinded to the therapy group to which the patient belonged. The patient, family member or person in charge was instructed not to comment on their management or activities they carried out, only to carry out the activities indicated by the evaluator during the review.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I: virtual reality activities (Experimental): The patient will practice the corresponding activities of the software indicated in the virtual reality equipment.
  Interventions: Behavioral: Virtual reality
- Group II: Modified Constraint-Induced Movement Therapy (Experimental): Patients will have the "healthy" upper limb fixed to the thorax with a sling and a horizontal shoulder immobilizer; The participants will practice physical and occupational therapy activities with the paretic upper limb.
  Interventions: Behavioral: Modified constraint-induced movement therapy
- Group III: Usual Physical and Occupational Therapy (Active Comparator): The participants will practice physical and occupational therapy activities that are usually provided in the Medical Unit, without any restrictions on the upper extremities.
  Interventions: Behavioral: Usual Physical and Occupational Therapy

INTERVENTIONS:
Behavioral: Virtual reality — The activities will be carried out with the Virtual Reality team, for 1 hour, twice a week, for 12 sessions (6 weeks). It will be indicated to repeat the activities at home, on similar equipment and with the same or similar software, at least 1 hour a day, at least 3 days a week.
  Arms: Group I: virtual reality activities
Behavioral: Modified constraint-induced movement therapy — Physical and occupational therapy activities will be carried out with the paretic upper limb, while the patient has the healthy upper limb "attached to the chest", for 1 hour, twice a week, for 12 sessions (6 weeks). It will be indicated to repeat the activities at home, 1 hour a day, at least 3 days a week. In addition, the participant will perform activities of daily living with the "free" paretic arm and the "fixed" healthy arm, for 5 hours a day.
  Arms: Group II: Modified Constraint-Induced Movement Therapy
Behavioral: Usual Physical and Occupational Therapy — The physical and occupational therapy activities that are usually practiced in the Medical Unit will be carried out for 1 hour, twice a week, for 12 sessions (6 weeks). It will be indicated to repeat the activities at home, for 1 hour a day, at least 3 days a week.
  Arms: Group III: Usual Physical and Occupational Therapy

SUMMARY:
The objective of this clinical trial is to measure the effect of Rehabilitation with Virtual Reality or Modified Constraint-Induced Movement Therapy on hemiparesis in patients with Cerebral Vascular Event.

The question to be answered is: What is the effect of different therapeutic modalities supported by Virtual Reality or Modified Constraint-Induced Movement Therapy compared with usual Physical and Occupational Therapy on motor recovery of paretic limbs in patients with Cerebrovascular Event?

The patients will carry out activities of:

* Virtual reality or
* Movement Restriction-Induction Therapy.

The investigators will compare the changes in the functionality of the paretic hemibody with a group undergoing regular physical and occupational therapy, as well as language and treatment-related satisfaction.

DETAILED DESCRIPTION:
Patients with diagnosis of cerebrovascular event (CVE) will be recruited upon arrival at the Medical Unit in the first appointment area; The diagnosis will be verified and an appointment will be made to the office of one of the researchers -rehabilitation specialist- (evaluator 1). During the appointment the purpose of the study will be explained and doubts will be clarified. All participants, whether accept or not, will receive the consultation that is normally provided to these patients and the information will be recorded in the medical record. If the subject does not accept, after the consultation, the appropriate management for the condition will be prescribed and a subsequent appointment will be made with another corresponding doctor to continue with the control.

If the subject agrees to participate, a clinical summary will be prepared, which will include demographic data, employment situation, the need for temporary disability for work and clinical data for the research file. The signature of the informed consent letter will also be requested. This physician 1 will assign the therapeutic modality using a table of random numbers to: Group 1. Therapy supported by virtual reality; Group 2. Modified Constraint-Induced Movement Therapy; o Group 3. Usual physical and occupational therapy. The activities corresponding to each group will be carried out during 2 sessions a week, of 1 hour each session, for 6 weeks.

An appointment will be made to be assessed by the second rehabilitation specialist (evaluator 2), who will remain blind to the treatment, and will measure the functionality of the thoracic and pelvic limbs with the different scales (Fugl-Meyer, Motor Index and Fine Clamp Test), including muscle tone, trophism, arcs of mobility, functionality of the limbs, as well as of the hand, coordination, balance and sensory aspects. These scales will be applied before (initial assessment -A.I.-), during (intermediate assessment -Int.A.- week 3, session 6) and after (final assessment -F.A. - week 6, session 12) of the different rehabilitation programs. During the same times, the Boston Aphasia Intensity scale and the Intrinsic Motivation Inventory will be applied by a neuropsychologist blinded to the treatment, for the evaluation of language and satisfaction, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients between 35 and 70 years of age and with a clinically and tomographically proven diagnosis of a cerebral vascular event in the territory of the middle cerebral artery.
* Patients with hemiparesis secondary to the cerebrovascular event
* Patients with a maximum Ashworth of 2 and Brunnstrom of minimum 4
* Patients with or without aphasia
* Patients with evolution between 1 to 3 months from hospital discharge of the cerebrovascular event
* Patients with cerebrovascular event of any sex
* Patients with vascular event without cognitive deficit
* Patients who agree to participate by signing an informed consent, by them or their family member or person in charge.

Exclusion Criteria:

* Patients who develop dementia or neurological-psychomotor complications during the study.
* Patients who present a new cerebrovascular event during the investigation
* Patients who do not complete at least 90% of the program
* Patients in whom a lack of family support or secondary gain is detected.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Estimated)
Dates: Start 2018-08-17 (Actual); Primary Completion 2024-08-21 (Actual); Study Completion 2024-08-21 (Estimated)

PRIMARY OUTCOMES:
Functionality and disability of the paretic hemibody due to evento vascular cerebral (CVE) to the 3 weeks of treatment. | Fugl-Meyer scale will be administered at week 3 of follow-up (just after completing 6 rehabilitation sessions).
  The motor functionality and disability of the paretic hemibody will be evaluated with Fugl-Meyer scale, it comprises 5 dominions y 113 total items that are scored on a 3 point ordinal scale (0= cannot perform, 1=perform partially, 2= perform fully).
  The individual scores are summed and the assessment can show a minimum value of 0 and a maximum value of 226 points, including 66 points for the upper extremity and 34 points for the lower extremity.
  A higher score represents better functionality of the hemibody (less disability).
Functionality and disability of the paretic hemibody due to cerebro vascular event (CVE) to the 6 weeks of treatment. | The Fugl-Meyer scale will be administered at week 6 of follow-up (just after completing the 12 rehabilitation sessions).
  The change in motor functionality and disability of the paretic hemibody will be evaluated with Fugl-Meyer scale, with 5 dominions y 113 total items that are scored on a 3 point ordinal scale (0= cannot perform, 1=perform partially, 2= perform fully).
  The individual scores are summed and the assessment can show a minimum value of 0 and a maximum value of 226 points, including 66 points for the upper extremity and 34 points for the lower extremity.
  Changes to higher score represents better functionality of the hemibody (less disability).
Independency of patient with hemiparesis secondary to cerebro vascular event (CVE) to the 3 weeks of treatment. | Motor Index scale will be administered at week 3 of follow-up (just after completing 6 therapy sessions).
  The motor functionality and independency of patient with paretic hemibody will be evaluated with motor index scale, it comprises 3 dominions and 5 items (two for upper limb, one to hand -grip-, and two to lower limb). In each domain can be obtained a minimum value of 0 and a maximum value of 33 points, and 1 point is added to the sum of all of them for the total qualification.
  A higher qualification represents a better ability to carry out activities of daily human life (greater independency).
Independency of patient with hemiparesis secondary to cerebro vascular event (CVE) to the 6 weeks of treatment. | The Motor Index scale will be administered at week 6 of follow-up (just after completing the 12 therapy sessions).
  The motor functionality and independency of patient with paretic hemibody will be evaluated with motor index scale, it comprises 3 dominions and 5 items (two for upper limb, one to hand -grip-, and two to lower limb). In each domain can be obtained a minimum value of 0 and a maximum value of 33 points, and 1 point is added to the sum of all of them for the total qualification.
  Changes to higher qualification represents a better ability to carry out activities of daily human life (greater independency).
Realization of the fine clamp of the plegia hand due to cerebro vascular event (CVE) to the 3 weeks of treatment. | Fine clamp test will be administered at week 3 of follow-up (just after completing 6 therapy sessions).
  The realization of grip of the plegia hand will be evaluated with the fine clamp test, it comprises three action for cubes take of size different (score: 0- inability to take the cube, 1- Grab with your whole hand, 2- Radial clamp or 3 finger clamp and 3- Forefinger thumb clamp). The total qualification has a minimum value of 0 and a maximum value of 9 points.
  A higher score represents a better performance of the clamp between the index finger and thumb of the paralyzed hand.
Realization of fine clamp of the plegia hand due to cerebro vascular event (CVE) to the 6 weeks of treatment. | Fine clamp test will be administered at week 6 of follow-up (just after completing 12 therapy sessions).
  The realization of grip of the plegia hand will be evaluated with the fine clamp test, it comprises three action for cubes take of size different (score: 0- inability to take the cube, 1- Grab with your whole hand, 2- Radial clamp or 3 finger clamp, and 3- Forefinger thumb clamp). The total qualification has a minimum value of 0 and a maximum value of 9 points.
  A higher score represents a better performance of the clamp between the index finger and thumb of the paralyzed hand.

SECONDARY OUTCOMES:
Level of aphasy to the 3 weeks of treatment. | Boston Aphasia Intensity scale will be administered at week 3 of follow-up (just after completing 6 rehabilitation sessions).
  The quality of language will be evaluated with the Boston Aphasia Intensity scale in patients after cerebro vascular event (CVE).
  In the Boston Aphasia Intensity scale the result has a minimum value of 0 and a maximum value of 5 points.
  A higher score represents a better language quality (less aphasy).
Level of aphasy to the 6 weeks of treatment. | Boston Aphasia Intensity scale will be administered at week 6 of follow-up (just after completing 12rehabilitation sessions).
  The quality of language will be evaluated with the Boston Aphasia Intensity scale in patients after cerebro vascular event (CVE).
  In the Boston Aphasia Intensity scale the result has a minimum value of 0 and a maximum value of 5 points.
  A higher score represents a better language quality (less aphasy).
Level of patient satisfaction with treatment to the 3 weeks of treatment. | Intrinsic Motivation inventory will be administered at week 3 of follow-up (just after completing 6 rehabilitation sessions).
  The satisfaction reported by the patient with the treatment received will be evaluated, with the Intrinsic Motivation inventory.
  In the Intrinsic Motivation inventory the result has a minimum value of 22 and a maximum value of 154 points. Score: from 1 (no satisfaction) to 7 (maximum satisfaction).
  A higher score represents a best level of satisfaction
Level of patient satisfaction with treatment to the 6 weeks of treatment. | Intrinsic Motivation inventory will be administered at week 6 of follow-up (just after completing 12 rehabilitation sessions).
  The satisfaction reported by the patient with the treatment received will be evaluated, with the Intrinsic Motivation inventory.
  In the Intrinsic Motivation inventory the result has a minimum value of 22 and a maximum value of 154 points. Score: from 1 (no satisfaction) to 7 (maximum satisfaction).
  A higher score represents a best level of satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: María del Carmen Rojas-Sosa, Doctorado, Principal Investigator — Instituto Mexicano del Seguro Social
Locations (1):
- Instituto Mexicano del Seguro Social, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-08-21): https://cdn.clinicaltrials.gov/large-docs/16/NCT05875116/Prot_SAP_ICF_000.pdf